CLINICAL TRIAL: NCT06023225
Title: Relationship Between Sex Hormones, Postoperative Pain and Opioid Use: the Role of Immune Factors
Brief Title: Sex Hormones, Postoperative Pain and Opioid Use
Acronym: SPO
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Hadas Nahman-Averbuch, Asst Prof of Anesthesiology, Washington University School of Medicine
Other Study IDs: 202210083
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postoperative patients: Pediatric female patients undergoing a surgical procedure
  Interventions: Behavioral: Pain; Behavioral: Opioid use

INTERVENTIONS:
Behavioral: Pain — Postoperative pain levels
Behavioral: Opioid use — Postoperative opioid use

SUMMARY:
Aim 1- To identify relationships between sex hormone levels and postoperative pain and opioid use.

Aim 2: To determine whether the effects of testosterone on postoperative pain and opioid use are mediated by immune factors

DETAILED DESCRIPTION:
After signing the consent and assent forms, participants and their parents/guardians will complete several surveys, including demographic, behavioral, pain, substance use and analgesic risk assessment measures, and developmental surveys. In addition, a blood sample (for hormonal and immune analyses) will be collected on the day of the surgery and/or postoperative. Surgery-related parameters including postoperative pain, and opioid type and doses during the hospital time will be collected.

In addition, before or after the surgery, patients and their parents/guardians will be interviewed. The interview will include questions about the surgery and about potential future study assessing the efficacy of sex hormone treatment on opioid use.

Longitudinal measures. At routine follow-up with the surgeons or after 1 week, 1 month, 3 months, and 6 months, study staff will contact patients to inquire about persistent pain (location, severity), and persistent opioid use. Based on previous studies, we estimate that ∼30% will have persistent postoperative pain, and ∼5% will have persistent opioid use.After signing the consent and assent forms, participants and their parents/guardians will complete several surveys, including demographic, behavioral, pain, substance use and analgesic risk assessment measures, and developmental surveys. In addition, a blood sample (for hormonal and immune analyses) will be collected on the day of the surgery and/or postoperative. Surgery-related parameters including postoperative pain, and opioid type and doses during the hospital time will be collected.

In addition, before or after the surgery, patients and their parents/guardians will be interviewed. The interview will include questions about the surgery and about potential future study assessing the efficacy of sex hormone treatment on opioid use.

Longitudinal measures. At routine follow-up with the surgeons or after 1 week, 1 month, 3 months, and 6 months, study staff will contact patients to inquire about persistent pain (location, severity), and persistent opioid use. Based on previous studies, we estimate that ∼30% will have persistent postoperative pain, and ∼5% will have persistent opioid use.

ELIGIBILITY:
Inclusion Criteria:

Pediatric female patients between the ages 11-16 undergoing an orthopedic (trauma and non-trauma) surgical procedure involving a long bone or joint, or the spine, English speaking

Exclusion Criteria:

Pregnancy; Diagnosis of chronic pain, Psychiatric, developmental or neurological disorders, Disorders that are associated with pubertal maturation (e.g., precocious puberty).

Ages: 11 Years to 16 Years | Sex: Female
Age Groups: Child
Study Population: Pediatric female patients between the ages 11-16 undergoing an orthopedic surgical procedure
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Sex hormone level of Testosterone | Baseline
Sex hormone level of estrogen | Baseline
Sex hormone level of progesterone | Baseline
Levels of IL-10 and IL-6 | Baseline
  Immune factors

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No